CLINICAL TRIAL: NCT06039930
Title: Tele-PROTECT Therapy: Effectiveness, Empowerment, and Implementation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York City Department for the Aging (Other); National Institute of Mental Health (NIMH) (NIH); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-12025491; R01MH132757 (NIH)
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Depression; Elder Abuse
Keywords: Elder Abuse; Depression; Mental Health
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The investigators will compare the effectiveness of the Tele- PROTECT Intervention against the Depression Education (DepEd) Intervention. To ensure rigor and reproducibility, Tele-PROTECT or DepEd will be offered to randomly assigned depressed elder abuse victims, and standard assessments will be conducted by trained raters blind to participant assignment and our hypotheses.
Who Masked: Outcomes Assessor
Masking Description: Standardized assessments will be conducted by trained raters blind to participant assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tele-PROTECT (Effectiveness Aim, Abuse Impact Aim) (Experimental): This group of participants will receive the Tele-PROTECT intervention, a behavioral intervention for depressed elder abuse (EA) victims designed to work in synergy with EA resolution services that provide safety planning, support services, and links to legal services.
  Interventions: Behavioral: Tele PROTECT
- Depression Education (DepEd) (Effectiveness Aim, Abuse Impact Aim) (Active Comparator): This group of participants will receive the Depression Education intervention, an intervention designed with active therapeutic ingredients (education, support, empathy) and designed to be what a good clinician providing education would do with an individual with depression.
  Interventions: Behavioral: Depression Education
- Stakeholder Groups (Implementation Aim) (No Intervention): To address the Implementation Aim of the study, investigators will conduct qualitative data via surveys, interviews, and focus groups. Qualitative data from NAPSA surveys, interviews, and focus groups will be analyzed to identify barriers and facilitators to the implementation of Tele-PROTECT in elder abuse agencies nation-wide using a mixed methods design with multiple stakeholder groups (e.g., EA directors, staff) in collaboration with the National Adult Protective Services Association (NAPSA).

INTERVENTIONS:
Behavioral: Tele PROTECT — Tele-PROTECT is a behavioral intervention delivered virtually over nine 45-minute sessions for depressed elder abuse (EA) victims. It is designed to work in synergy with EA resolution services that provide safety planning, support services, and links to legal services.
  Other Names: PROTECT
  Arms: Tele-PROTECT (Effectiveness Aim, Abuse Impact Aim)
Behavioral: Depression Education — DepEd is designed as an intervention delivered virtually over nine 45-minute sessions with active therapeutic ingredients (education, support, empathy). It is designed to be what a good clinician providing education would do with an individual with depression.
  Other Names: DepEd
  Arms: Depression Education (DepEd) (Effectiveness Aim, Abuse Impact Aim)

SUMMARY:
The purpose of this randomized trial is to conduct a fully powered effectiveness trial of video-delivered PROTECT (Tele-PROTECT) compared to a video-delivered depression education (DepEd) control condition to be delivered to 140 English- and Spanish-speaking NYC elder abuse victims. Investigators hypothesize three main aims:

1. Effectiveness Aim: Tele-PROTECT participants will have significantly greater and clinically meaningful reductions in depression when compared to the DepEd control;
2. Abuse Impact Aim: Tele-PROTECT participants will demonstrate greater safety related empowerment compared to DepEd control, which can help participants take steps to reduce risk;
3. Implementation Aim: Stakeholders' views of the factors impacting the implementation of Tele-PROTECT based on characteristics of the intervention, agency setting, and population served will contribute to a national dissemination of Tele-PROTECT

Participants will

* Receive 9 weeks of tele health psychotherapy delivered by a Master's level mental health clinician from the Weill Cornell Medicine research team. Participants will be assigned to "Tele-PROTECT" or "DepEd" psychotherapy randomly.
* Participate in one baseline assessment and four follow-up assessments at weeks 3, 6, 9, and 12 administered by a trained member of the research team.

DETAILED DESCRIPTION:
The WHO estimates that 1 in 6 older adults have experienced elder abuse in the past year with rates in the community increasing by as much as 83.6% during the pandemic. Elder abuse (EA) takes a serious physical and emotional toll on older adults, including premature mortality, physical injuries and financial losses. EA victims in NYC are more likely to be women than men, and more likely to be women of color.

Previous work by the investigators has demonstrated that 1/3 of victims have clinically significant depressive symptoms. Abused older adults with depression have higher rates of mortality and suicidal ideation. Depression is an additional barrier to implementing safety steps to reduce victimization. PRoviding Options To Elderly Clients Together (PROTECT) is a behavioral intervention for depressed elder abuse victims. It is the only manualized therapy for depressed elder abuse victims designed to be integrated with elder abuse services. It is aligned with the NIMH Strategic Plan "to deliver high quality, impactful research and promote translation of such research into clinical practice" and to serve "underrepresented and underserved communities."

The investigators developed PROTECT to work in synergy with abuse resolution services. PROTECT reduces depression by increasing engagement in pleasurable and rewarding activities and taking steps towards goals to reduce threat. PROTECT has been designed in an iterative process with partners at the New York City (NYC) Dept. for the Aging (DFTA). In the investigators' pilot randomized controlled trial, PROTECT showed an increase in behavioral activation (BADS) and significantly decreased depression as compared to a referral control condition. PROTECT has been adopted by DFTA (Community PROTECT) to increase its use.

In collaboration with partners at DFTA and five NYC elder abuse agencies, the investigators propose a fully powered effectiveness trial of video-delivered PROTECT (Tele-PROTECT) compared to a video- delivered depression education (DepEd) control condition to be delivered to 140 English- and Spanish- speaking NYC elder abuse victims. In partnership with a national elder abuse organization (NAPSA), and using the CFIR, the investigators will examine factors that could affect future implementation of Tele-PROTECT nationally.

ELIGIBILITY:
Inclusion Criteria:

* ≥60 years of age
* Capacity to consent (per elder abuse staff)
* Depression, i.e., PHQ-9≥10 (by elder abuse staff), represents mild to moderate severity of depression and has a sensitivity of 88% and a specificity of 88% for major depression
* Need for elder abuse services as verified by the elder abuse case worker.

Exclusion Criteria:

* Active suicidal ideation (MADRS item 10 ≥4)
* Inability to speak English or Spanish
* Axis 1 DSM-5 diagnoses other than unipolar depression or comorbid generalized anxiety disorder (by SCID)
* Mini-MOCA less than 11
* Severe or life-threatening medical illness
* Elder abuse emergency and or referral out of elder abuse agency.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | Assessed at baseline and week three of treatment
  The Montgomery Asberg Depression Rating Scale (MADRS) is a 10-item scale that assesses depression severity. Scores range from 0 to 60, with a score of 0 indicating no depressive symptoms present and a score of 60 indicating severe depression. Scores will be used to assess depression severity outcome and evaluate the impact of interventions in line with the Effectiveness Aim.
Montgomery Asberg Depression Rating Scale (MADRS) | Assessed baseline and week six of treatment
  The Montgomery Asberg Depression Rating Scale (MADRS) is a 10-item scale that assesses depression severity. Scores range from 0 to 60, with a score of 0 indicating no depressive symptoms present and a score of 60 indicating severe depression. Scores will be used to assess depression severity outcome and evaluate the impact of interventions in line with the Effectiveness Aim.
Montgomery Asberg Depression Rating Scale (MADRS) | Assessed baseline and week nine of treatment
  The Montgomery Asberg Depression Rating Scale (MADRS) is a 10-item scale that assesses depression severity. Scores range from 0 to 60, with a score of 0 indicating no depressive symptoms present and a score of 60 indicating severe depression. Scores will be used to assess depression severity outcome and evaluate the impact of interventions in line with the Effectiveness Aim.
Montgomery Asberg Depression Rating Scale (MADRS) | Assessed baseline and 3 weeks after treatment end, approximately 12 weeks from enrollment
  The Montgomery Asberg Depression Rating Scale (MADRS) is a 10-item scale that assesses depression severity. Scores range from 0 to 60, with a score of 0 indicating no depressive symptoms present and a score of 60 indicating severe depression. Scores will be used to assess depression severity outcome and evaluate the impact of interventions in line with the Effectiveness Aim.
Measure Of Victim Empowerment Related to Safety (MOVERS) Scale | Assessed at baseline and week three of treatment
  The MOVERS a 13-item scale assesses the presence of a set of safety-related goals, the ability to accomplish them, and victims' sense that others can and will assist them as needed. Scores range from 13 to 65 with higher scores indicating a greater degree of empowerment related to safety. The MOVERS serves to measure the Abuse Impact Aim.
Measure Of Victim Empowerment Related to Safety (MOVERS) Scale | Assessed at baseline and week six of treatment
  The MOVERS a 13-item scale assesses the presence of a set of safety-related goals, the ability to accomplish them, and victims' sense that others can and will assist them as needed. Scores range from 13 to 65 with higher scores indicating a greater degree of empowerment related to safety. The MOVERS serves to measure the Abuse Impact Aim.
Measure Of Victim Empowerment Related to Safety (MOVERS) Scale | Assessed at baseline and week nine of treatment
  The MOVERS a 13-item scale assesses the presence of a set of safety-related goals, the ability to accomplish them, and victims' sense that others can and will assist them as needed. Scores range from 13 to 65 with higher scores indicating a greater degree of empowerment related to safety. The MOVERS serves to measure the Abuse Impact Aim.
Measure Of Victim Empowerment Related to Safety (MOVERS) Scale | Assessed baseline and 3 weeks after treatment end, approximately 12 weeks from enrollment
  The MOVERS a 13-item scale assesses the presence of a set of safety-related goals, the ability to accomplish them, and victims' sense that others can and will assist them as needed. Scores range from 13 to 65 with higher scores indicating a greater degree of empowerment related to safety. The MOVERS serves to measure the Abuse Impact Aim.

SECONDARY OUTCOMES:
2 item survey assessing agency access to mental health services | Year 3 of study duration
  In line with the Implementation Aim, agency access to mental health services will be assessed with a 2 item survey evaluating the method by which agencies access mental health services for clients (response options: the agency provides services, outside agency referral, no access) and mental health service availability (response options: 0=not at all available; 5=very available).
Organizational Change Manager (OCM) | Year 3 of study duration
  In line with the Implementation Aim, subscales of the Organizational Change Manager (OCM) scale will be used to assess: Relative advantage (3 items), Tension for change (3 items), and Goals and feedback (2 items). Items are rated on a five-point scale with higher scores indicating greater likelihood of implementation. Barriers/facilitators to mental health service provision across the Consolidated Framework for Implementation Research (CFIR) domains will be assessed with this and other measures.
The Organizational Readiness to Change Assessments (ORCA) | Year 3 of study duration
  In line with the Implementation Aim, the ORCA will be used to assess client needs and resources (3 items). ORCA is a reliable and valid measure of organization readiness to implement change and barriers of that change. Each item is rated on a five-point scale with higher scores indicating greater organizational readiness for change

CONTACTS AND LOCATIONS:
Overall Officials: Jo Anne Sirey, Ph.D, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The Center will share its data via the NIMH Data Archive (NDA). Our resource sharing plan is formulated in accordance with the NDA Data Sharing Terms and Conditions. Further, the Center will use NDA technologies to submit data in accordance with the NDA Data Sharing Terms and Conditions. This project will share data comparing the effectiveness of the Tele-PROTECT Intervention against the Depression Education (DepEd) Intervention. Investigators will comply with NIMH's procedures for data deposition into NDCT, and will let NDCT policies dictate the timetable upon which and avenues through which others will be allowed to access those data. Investigators will make the dataset available to other researchers after the main results have been published. Investigators will de- identify the data in the final datasets prior to release for sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Per NIMH guidelines
Access Criteria: To ensure data and participant security, investigators will make the data available to users only under a data-sharing agreement. All users will make a direct request to the Principal Investigator with a proposal of hypotheses, variables needed to test these hypotheses, and plans for dissemination of findings. All users will indicate in a signed document: (1) a commitment to using the data only for research purposes; (2) a plan for securing the data; (3) an agreement to either destroying or returning the data once analyses are completed; and (4) an agreement to not share data with other users and to direct all such requests to the Principal Investigator.